CLINICAL TRIAL: NCT06440252
Title: The Effectiveness of a Grape Seed Extract on Circulatory Measures in Healthy Adults: a Randomised, Double-blind, Placebo-controlled Crossover Study
Brief Title: Effectiveness of a Grape Seed Extract on Circulatory Measures in Healthy Adults
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ALVCIR
Record Dates: First submitted 2024-05-17; First posted 2024-06-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Circulatory; Change
MeSH Terms: interventions — Grape Seed Extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grape Seed Extract (Active Comparator): Grape seed extract 600mg per day - 1 capsule per day
  Interventions: Drug: Grape Seed Extract
- Maltodextrin (Placebo Comparator): Maltodextrin - 1 capsule per day
  Interventions: Drug: Maltodextrin

INTERVENTIONS:
Drug: Grape Seed Extract — One daily dose of 1 capsule containing 600mg grape seed extract
  Arms: Grape Seed Extract
Drug: Maltodextrin — One daily dose of 1 capsule
  Arms: Maltodextrin

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2 arm crossover study conducted over 11 weeks, with participants randomised to a product for 4 weeks, followed by a 3-week washout period before completing the second product for 4 weeks, to study the effectiveness of a grape seed extract on circulatory measures in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults 25 years or older
* Generally healthy
* BMI 18 - 35kg/m2
* Able to provide informed consent
* Have prehypertensive blood pressure (systolic 120-139 mmHg and/or diastolic 80-89 mmHg)
* Agree to not change current diet and/or exercise frequency or intensity during entire study period
* Agree to not participate in another clinical trial while enrolled in this trial

Exclusion Criteria:

* Those with a history of myocardial infarction, angina or bleeding disorders
* Those who have uncontrolled thyroid diseases
* Currently taking dietary supplements for circulation (e.g. fatty acids, CoQ10, L-arginine, red ginseng, ginseng, natto, ginkgo) or use of these in the last 1 month
* Currently taking inflammation or circulatory associated medications (e.g. Pentoxifylline and vasodilators like nitroglycerin) or use of these in the last 1 month
* Currently taking statins medication including atorvastatin (e.g. Lipitor, Lorstat), fluvastatin (e.g. Lescol or Vastin), pravastatin (e.g. Pravachol, Cholstat), rosuvastatin (e.g. Cavstat, Crestor) or simvastatin (e,g, Lipex, Zocor, Zimstat).
* Currently taking Coumadin, Marevan (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy, or substrates of P-glycoprotein including (but not limited to) calcium channel blockers, cyclosporin, digoxin, erythromycin and protease inhibitors(1).
* Have a serious illness(2) e.g. mood disorders such as bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Have an unstable illness(3) (i.e., changing medication/treatment)
* Malignancy or treatment for malignancy within the previous 2 years (this excludes non-melanoma (e.g. BCC and SCC) skin cancers not requiring radiation or chemotherapy)
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in active or placebo formula
* Pregnant or lactating woman or women trying to conceive
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion
* Participated in another trial in the past 1 month

  1. Any participant that begins taking antiplatelet medication during the trial will be excluded from the study
  2. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
  3. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Diastolic blood pressure (arm) | Baseline, week 4, week 8, week 11
  Change in Diastolic blood pressure (arm) as measured by blood pressure machine

SECONDARY OUTCOMES:
Change in Systolic blood pressure (arm) | Baseline, week 4, week 8, week 11
  Change in Systolic blood pressure (arm) as measured by blood pressure machine
Change in Peripheral systolic and diastolic blood pressure (leg) | Baseline, week 4, week 8, week 11
  Change in Peripheral systolic and diastolic blood pressure (leg) as measured by blood pressure machine
Change in HGB | Baseline, week 4, week 8, week 11
  Change in HGB as measured by FBC via blood test
Change in WBC | Baseline, week 4, week 8, week 11
  Change in WBC as measured by FBC via blood test
Change in RBC | Baseline, week 4, week 8, week 11
  Change in RBC as measured by FBC via blood test
Change in Platelet Aggregation | Baseline, week 4, week 8, week 11
  Change in Platelet Aggregation as measured by FBC via blood test
Change in (endothelial nitric oxide synthase) eNOS | Baseline, week 4, week 8, week 11
  Change in eNOS as measured via blood test
Change in endogenous nitric oxide (NO) | Baseline, week 4, week 8, week 11
  Change in NO as measured via blood test
Change in Tibial artery structure | Baseline, week 4, week 8, week 11
  Change in Tibial artery structure via Laser Doppler Flowmetry
Change in blood flow of the right leg | Baseline, week 4, week 8, week 11
  Change in blood flow of the right leg via Laser Doppler Flowmetry
Change in oxygen saturation | Baseline, week 4, week 8, week 11
  Change in oxygen saturation as measured by pulse oximeter
Change in resting pulse rate | Baseline, week 4, week 8, week 11
  Change in resting pulse rate as digital blood pressure and resting pulse rate machine
Change in weight | Baseline, week 4, week 8, week 11
  Change in weight as measure by digital scales
Change in Body Mass Index (BMI) | Baseline, week 4, week 8, week 11
  Change in BMI as measured by weight and height calculation
Change in waist and hip circumference | Baseline, week 4, week 8, week 11
  Change in waist and hip circumference as measured by tape measure
Change in 36-Item Short Form Health Survey (SF-36) | Baseline, week 4, week 8, week 11
  Change in 36-Item Short Form Health Survey (SF-36) as self-reported
Change in E/LFT | Baseline, week 4, week 8, week 11
  Change in E/LFT as measured via blood test
Change in triglycerides | Baseline, week 4, week 8, week 11
  Change in triglycerides as measured via blood test
Change in cholesterol | Baseline, week 4, week 8, week 11
  Change in cholesterol as measured via blood test
Change in blood glucose | Baseline, week 4, week 8, week 11
  Change in blood glucose as measured via blood test
Change in adverse events | Baseline, week 4, week 8, week 11
  Change in adverse events as reported by participant

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Rao, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia